CLINICAL TRIAL: NCT00861640
Title: The Comparison of Oral Rabeprazole vs. Intravenous Omeprazole in the Treatment of Patients With Mild to Moderate Nonvariceal Upper Gastrointestinal Bleeding
Brief Title: Comparison of Oral Rabeprazole vs. iv Omeprazole in Mild to Moderate Nonvariceal Upper Gastrointestinal Bleeding
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Kaohsiung Medical University (Other)
Responsible Party: Chien-Yu Lu, Kaohsiung Medicial University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMUH-IRB-970338
Record Dates: First submitted 2009-03-11; First posted 2009-03-13 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Nonvariceal Upper Gastrointestinal Bleeding
Keywords: rabeprazole; omeprazole; upper gastrointestinal bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Omeprazole; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous Omeprazole (Experimental): 100 cases of Intravenous Omeprazole
  Interventions: Drug: Intravenous Omeprazole
- Oral Rabeprazole (Experimental): 100 cases of oral rabeprazole
  Interventions: Drug: Oral Rabeprazole

INTERVENTIONS:
Drug: Intravenous Omeprazole — Intravenous Omeprazole 1amp qd (every day)
  Other Names: iv losec
  Arms: Intravenous Omeprazole
Drug: Oral Rabeprazole — Oral Rabeprazole 1 bid
  Other Names: pariet
  Arms: Oral Rabeprazole

SUMMARY:
Introduction: Proton pump inhibitor (PPI) is the drug of choice used in patients with non-variceal upper gastrointestinal tract bleeding (UGIB). Intravenous (IV) PPI is more commonly used than oral form when overt bleeding occurs. Previous study has revealed that oral rabeprazole and IV omeprazole achieved similar intragastric pH elevation. It's probable that oral form and IV PPI provide equal efficacy in treating mild to moderate UGIB patients.

Aim: This study aims to compare the effect of three-day oral rabeprazole and iv omeprazole on bleeding control in patients with mild to moderate non-variceal UGIB.

Patients and methods: All patients presented with black to tarry stool passage or hematemesis and visited our ER will be evaluated to recruit into this study. They will receive regular vital sign monitoring, laboratory study and nasogastric tube insertion with gastric fluid aspiration. Esophagogastroendoscopy and hemostatic procedure if need will be performed within 12 hours. Those confirmed to have non-variceal UGIB, stable vital signs and agree to participate into this study will be randomized into two groups receiving either oral rabeprazole (20mg bid) or iv omeprazole (40mg qd) for three days. The presence of recurrent bleeding within three days, in-hospital complication and duration of hospital stay will be recorded and analyzed.

Expected results: At the end of this study, we will be able to determine whether patients treated with oral rabeprazole and iv omeprazole have similar re-bleeding or complication rates and hospitalization days.

DETAILED DESCRIPTION:
Proton pump inhibitor (PPI) is the drug of choice used in patients with non-variceal upper gastrointestinal tract bleeding (UGIB). Intravenous (IV) PPI is more commonly used than oral form when overt bleeding occurs. Previous study has revealed that oral rabeprazole and IV omeprazole achieved similar intragastric pH elevation. It's probable that oral form and IV PPI provide equal efficacy in treating mild to moderate UGIB patients.

This study aims to compare the effect of three-day oral rabeprazole and iv omeprazole on bleeding control in patients with mild to moderate non-variceal UGIB. The expected numbers of intravenous and oral PPI were 100 respectively.

All patients presented with black to tarry stool passage or hematemesis and visited our ER will be evaluated to recruit into this study. They will receive regular vital sign monitoring, laboratory study and nasogastric tube insertion with gastric fluid aspiration. Esophagogastroendoscopy and hemostatic procedure if need will be performed within 12 hours. Those confirmed to have non-variceal UGIB, stable vital signs and agree to participate into this study will be randomized into two groups receiving either oral rabeprazole (20mg bid) or iv omeprazole (40mg qd) for three days. The presence of recurrent bleeding within three days, in-hospital complication and duration of hospital stay will be recorded and analyzed.

At the end of this study, we will be able to determine whether patients treated with oral rabeprazole and iv pantoprazole have similar re-bleeding or complication rates and hospitalization days.

ELIGIBILITY:
Inclusion Criteria:

* moderate to mild upper gastrointestinal peptic ulcer bleeding

Exclusion Criteria:

* shock
* liver cirrhosis
* uremia
* severe UGI bleeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
This study aims to compare the effect of three-day oral rabeprazole and iv omeprazole on bleeding control in patients with mild to moderate non-variceal UGIB. | one year later

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Yu Lu, MD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan